CLINICAL TRIAL: NCT00953823
Title: The Prevalence of Thiamin Deficiency in Ambulatory Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, mary keith, Coordinator of Nutrition and Dietetic Education/Research, Unity Health Toronto
Other Study IDs: REB 09-031
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Heart Failure
Keywords: Thiamin supplementation; Thiamin deficiency; Heart failure; Heart function; Vitamin B1 supplementation
MeSH Terms: conditions — Heart Failure; Beriberi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood test
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with heart failure are at an increased risk for thiamin deficiency (TD), for many reasons such as malnutrition and the use of diuretic drugs. Thiamin is a B vitamin that plays an important role in the production of energy in body. Therefore, low levels of thiamin may limit the amount of energy available for the heart to pump blood. Recent thiamin supplementation trials have demonstrated significant improvements in heart function. However, while clinically important, the results of these studies are limited by their small sample sizes, indirect measurement of thiamin status and reliance on hospitalized patients. Therefore, the investigators' goal is to determine the prevalence of thiamin deficiency in ambulatory patients with heart failure by direct measurement of thiamin in red blood cells.

DETAILED DESCRIPTION:
Thiamin is a water-soluble B-complex vitamin which is supplied primarily from cereals and enriched grains in the ordinary diet. The majority of absorbed thiamin combines with ATP in the body to form thiamin pyrophosphate (TPP). TPP is a coenzyme which is involved in a number of energy production reactions in the body (metabolism of carbohydrates and some amino acids) . Therefore, theoretically, TD reduces the release of metabolic energy in the tissues . The adverse effects of TD include biventricular myocardial failure, tachycardia, peripheral edema, and retention of sodium which occurs as a result of heart failure . Therefore, our assumption is that TD in CHF patients may result in depletion of cellular energy and subsequently impair cardiac function. Previous studies done on CHF patients with TD found that thiamin supplementation was associated with improvement in heart contractility.

Patients with heart failure are at an increased risk for TD, for many reasons such as malnutrition, anorexia and the use of diuretic drugs, such as furosemide. Several studies have demonstrated a high prevalence of TD in hospitalized patients with heart failure, ranging from 13 % to 91% depending on the population studied. This wide variation is due to differences in the underlying nutrition status of subjects, the concurrent use of medications including loop diuretics, the severity of disease, and the measurement technique used for the assessment of thiamin status. These studies however, while clinically important, are limited by their small sample size and indirect measurement of thiamin status. Also, these studies have focused exclusively on the hospitalized patients, whereas ambulatory HF patients have received little attention.

Therefore, our primary objective to conduct a prospective, cross-sectional study to investigate the prevalence of thiamin deficiency in a large group of ambulatory patients with heart failure using High-Performance Liquid Chromatography (HPLC). This method has many advantages including its high level of recovery (102% on average), high intra- and inter-day precisions within 5-9%, as well as having a considerably low elution time of 15 min.

Our secondary objective is to conduct a trial using oral thiamin supplements alone in three practical doses in order to estimate the minimum dose of oral thiamin required to effectively replete tissue stores. We also hypothesize that oral thiamin supplementation will reduce neurohormonal stimulation (NE, BNP,as well as oxidative stress(F2-Isoprostanes).

Therefore,this study will provide critical data on the prevalence of TD in ambulatory patients with HF as well as defining what factors are predictive of TD in this population. Furthermore, this study will determine an effective dose of oral thiamin supplementation that will restore red blood cell thiamin levels. Determining an effective dose will not only justify our choice of thiamin supplementation in future studies but will guide clinicians in recommending thiamin supplementation to their patients with heart failure in the community.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the primary diagnosis of ischemic, dilated, idiopathic or valvular HF characterized by an ejection fraction of < 45% (echocardiography or radionuclide scan)
* Patients with NYHA class I-IV symptoms

Exclusion Criteria:

* Patients who are unable or unwilling to provide informed consent
* Patients with any concurrent condition which would result in TD, namely, gastrointestinal disorders (Crohn's disease, ulcerative colitis), liver disease, prolonged diarrhoeal disease, dialysis, prolonged fever, infection or renal failure
* Patients who are rapidly deteriorating, who are not on a stable medication regimen (≥ 2 months) or have been hospitalized for acute decompensated HF in the last 2 months
* Patients who are on experimental medications
* Patients who consume excessive alcohol (> 3 drinks per day), have a documented history of alcoholism or have documented alcoholic cardiomyopathy
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology Clinic (St Michael's Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of Thiamin deficiency as determined by Erythrocyte thiamin pyrophosphate (TPP) measured using a direct HPLC technique | baseline

SECONDARY OUTCOMES:
Eligible patients will be randomized to one of three commercially available doses of oral thiamin hydrochloride; 50 mg QD, 50 mg BID and 100 mg BID. They will take the supplements for 2 weeks. | baseline to after two weeks of supplementation
Plasma samples will be analyzed for the plasma levels of NE, BNP, F2-isoprostanes | baseline and after supplementation
Urinary excretion of thiamin following the 2 week supplementation period. | by the end of two-week supplementation period

CONTACTS AND LOCATIONS:
Overall Officials: Mary Keith, PhD, RD, Principal Investigator — Unity Health Toronto; Andrew Yan, MD, Principal Investigator — Cardiologist, St. Michael's Hospital; Abdul Al-Hesayen, MD, Principal Investigator — Cardiologist, St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada